CLINICAL TRIAL: NCT05297201
Title: Phase II, Double Blind, Randomized, Placebo Controlled, Parallel Group, Trial to Explore the Potential Anti-dyskinetic Properties of CPL500036 (PDE10A Inhibitor) in Patients with Parkinson's Disease Suffering from Levodopa Induced Dyskinesia
Brief Title: Efficacy, Safety and Pharmacokinetic Study of CPL500036 in Patients with Levodopa Induced Dyskinesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celon Pharma SA (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03PDE2020
Record Dates: First submitted 2022-02-17; First posted 2022-03-28 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease; Dyskinesia, Medication-Induced
Keywords: Parkinson's; Levodopa induced dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesia, Drug-Induced

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CPL500036 low dose (Experimental): Patients will receive 20 mg of CPL500036 administered once daily for 28-days treatment period.
  Interventions: Drug: CPL500036 - low dose
- CPL500036 high dose (Experimental): Patients will receive 40 mg of CPL500036 administered once daily for 28-days treatment period.
  Interventions: Drug: CPL500036 - high dose
- Placebo (Placebo Comparator): Patients will receive placebo administered once daily for 28-days treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CPL500036 - low dose — CPL500036 will be given orally. Each patient is to take 2 capsules with active substance and 2 capsules of placebo daily.
  Arms: CPL500036 low dose
Drug: CPL500036 - high dose — CPL500036 will be given orally. Each patient is to take 4 capsules with active substance daily.
  Arms: CPL500036 high dose
Drug: Placebo — Placebo will be given orally. Each patient is to take 4 capsules of placebo daily.
  Arms: Placebo

SUMMARY:
The aim of the study is to determine potential anti-dyskinetic properties of CPL500036 (PDE10A inhibitor) in Parkinson disease patients suffering from levodopa Induced dyskinesia. The study is to determine the efficacy and dose response of two CPL500036 doses, compared with placebo.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, parallel-group, dose ranging study, to explore the efficacy, safety, tolerability and pharmacokinetic (PK) of low and high dose of CPL500036 an phosphodiesterase 10A (PDE10A) inhibitor in Parkinson's disease patients with levodopa induced dyskinesia (LID) when administered for 28 days. The study will be conducted at multiple Clinical Sites. Approximately 108 patients will be randomized at 1:1:1 ratio to receive low or high dose of CPL500036 or placebo in a blinded manner, once daily for 28 days (Day 1 to Day 28). The study will comprise of Screening, Baseline (a 4-day in-house period), a Treatment Period and a Follow-Up Period. The patients will be discharged from clinical units during the Treatment Period. Approximately 30% of the patients (11 patients in each of the 3 treatment groups) will undergo extensive PK blood sampling during the Treatment Period and the remaining 70% of the patients will undergo sparse PK blood sampling. Patients from extensive PK blood sampling will be discharged from the Clinical Site on Day 8 and Day 1 for patients from sparse PK blood sampling group respectively.

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated written informed consent.
2. Male or female patient aged between 50 and 80, diagnosed of idiopathic Parkinson's disease according to the United Kingdom Parkinson's Disease Society Brain Bank Clinical Diagnosis Criteria.
3. The patient is on stable dose of Levodopa.
4. Other anti-PD medications are allowed if dosing is optimized and stably used.
5. The patient is has been treated with Levodopa and is suffering from temporally predictable peak-dose LID.
6. Patient declare that dyskinesia is problematic or disabling.
7. Score of dyskinesia is at least 2 on part IV, item 4.2 (of the MDS-UPDRS at Screening and on Day -1).
8. Patient with Hoehn-Yahr stages 2 to 4 (in OFF stage).
9. Female patient is not pregnant (at Screening and Day -1), not breastfeeding and at least 1 of the following conditions applies: (i) woman of non-childbearing potential; (ii) woman of childbearing potential, using contraceptive methods during the Treatment Period and for at least 28 days after the last dose of the study drug.

   The following are acceptable contraceptive methods: bilateral tubal occlusion, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices and copper intrauterine devices, male or female condom with spermicide; and cap, diaphragm or sponge with spermicide.
10. Male patient must agree to use a barrier method of contraceptive for at least 90 days after the last dose of the study drug.
11. Patient agrees to blood sample collection for DNA analysis.

Exclusion criteria:

1. The patient has (suspected) atypical Parkinson's disease.
2. The patient has a history of neurosurgical intervention because of Parkinson's disease.
3. Patient has unstable medical status which may impact the ability of the patients to participate or potentially confound the study result.
4. Patient has a history of psychotic event induced by anti-PD treatments or impulse control disorder.
5. The patient has any moderate or severe neuromuscular, locomotor disease, that interfere with the study scoring.
6. The Patient has a history of severe head injury, stroke or any diagnosis of significant nervous system disease.
7. Patient has a history of substance abuse or alcohol abuse within 12 months prior to Screening.
8. The patient is pregnant or lactating or intending to become pregnant or intending to donate ova.
9. Patient has a history of neuroleptic malignant syndrome, or known personality disorder, or other psychiatric disorder that, in the opinion of the Investigator, would interfere with participation in the study.
10. Patient with the presence of cognitive impairment evidenced by a Mini-Mental State Exam (MMSE) of less than 19.
11. Patients is considered by the Investigator to be at imminent risk of suicide or injury to self or others.
12. Patients has any existing or previous history of cancer or has newly diagnosed diabetes.
13. Patient has abnormal ECG that, in the opinion of the Investigator, increases the risks associated with participating in the study.
14. Patient has abnormal QT interval, history of unexplained syncope or known family history of sudden death due to QT abnormality.
15. The patient has any laboratory values outside the normal range that are considered by Investigator to be clinically significant at Screening.
16. Patient participated in another interventional clinical study with an IMP

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total UDysRS score at Week 4. | Day -1, Day 28
  Determination of the effect of low and high dose of CPL500036 compared to placebo, on the reduction of dyskinesia based on Unified Dyskinesia Rating Scale (UDysRS). The UDysRR scale is used to measure dyskinesia in Parkinson disease. Within a single scale, rater is to evaluate patient perceptions, time factors, anatomical distribution, objective impairment, severity, and disability which are accordingly divided into Part 1, Part 2, Part 3 and Part 4 of the UDysRS scale, respectively.

SECONDARY OUTCOMES:
Change from baseline in UDysRS objective sub-scale scores Part 3 and 4. | Day -1, Week 1, 2, 3 and 4
  Determination of the effect of low and high dose of CPL500036 compared to placebo, on the reduction of dyskinesia based on Unified Dyskinesia Rating Scale (UDysRS). The UDysRR scale is used to measure dyskinesia in Parkinson disease. Within a single scale, rater is to evaluate patient perceptions, time factors, anatomical distribution, objective impairment, severity, and disability which are accordingly divided into Part 1, Part 2, Part 3 and Part 4 of the UDysRS scale, respectively.
Change from baseline in MDS-UPDRS total score at Week 4 | Day -1, Day 28
  Determination of the effect of low and high dose of CPL500036 compared to placebo using Movement Disorders Society (MDS) Modified Unified Parkinson's Disease Rating Scale (MDS-UPDRS). MDS-UPDRS is use to measure the severity and progression of Parkinson disease (PD). The MDS-UPDRS scale contain 4 parts that captures essential features of Parkinson's disease. Within a single scale, rater is to evaluate non-motor (Part 1) and motor (Part 2) experience of daily living, motor examination (Part III) and motor complications (Part IV).
Change from baseline in MDS-UPDRS Part 4/A scores at Week 4 | Day -1, Day 28
  Determination of the effect of low and high dose of CPL500036 compared to placebo using Movement Disorders Society (MDS) Modified Unified Parkinson's Disease Rating Scale (MDS-UPDRS). MDS-UPDRS is use to measure the severity and progression of Parkinson disease (PD). The MDS-UPDRS scale contain 4 parts that captures essential features of Parkinson's disease. Within a single scale, rater is to evaluate non-motor (Part 1) and motor (Part 2) experience of daily living, motor examination (Part III) and motor complications (Part IV).
Change from baseline in Hauser Subject Diary data in ON time with and without dyskinesia or with non-troublesome dyskinesia. | up to 6 weeks
  The Hauser Diary is use to monitor motor fluctuation. Patients are asked to characterize their prevailing motor states in 30-minute intervals.
Adverse events assessment | up to 6 weeks
  Number of all of adverse events will be assessed.
Cmax - maximum CPL500036 plasma concentration | up to 24 hours post administration on Day 1 and Day 7
  The maximum concentration of the CPL500036 compound in plasma after IMP administration, obtained directly from the measured concentrations.
Tmax - time to reach maximum CPL500036 concentration | up to 24 hours post administration on Day 1 and Day 7
  The Tmax is time to reach the maximum plasma concentration (Cmax), obtained directly from the actual sampling times.
AUC(0-24) - area under the plasma concentration - time curve from time 0 to 24 hours after IMP administration for CPL500036 | up to 24 hours post administration on Day 1 and Day 7
  The AUC(0-24) is a measure of total plasma exposure to the drug from time point zero to 24 hours after IMP administration.
AUC(0-inf) - area under the plasma concentration - time curve from time 0 to infinity time for CPL500036 | up to 24 hours post administration on Day 1 and Day 7
  The AUC(0-inf) is a measure of total plasma exposure to the drug from time point zero extrapolated to infinity.
Kel - terminal elimination rate constant | up to 24 hours post administration on Day 1 and Day 7
  Kel is to be estimated via linear regression of time versus log of concentration.
Apparent terminal elimination half-life (T1/2) for CPL500036 compound | up to 24 hours post administration on Day 1 and Day 7
  T1/2 is to be calculated as 0.693/Kel.
Apparent clearance (CL/F) for CPL500036 compound | up to 24 hours post administration on Day 1 and Day 7
  Apparent clearance is to be calculated as Dose/AUC(inf)
Apparent volume of distribution during the terminal phase (Vz/F) for CPL500036 compound | up to 24 hours post administration on Day 1 and Day 7
  Apparent volume of distribution is to be calculated as (CL/F)/ Kel
C(trough) - CPL500036 concentration before dosing | Day 1 and Day 7
  The concentration of CPL500036 on day before product administration.
Change from baseline in inflammatory cytokines level at Week 4 | Day 1, Day 28
  Determination of the effect of low and high dose of CPL500036 compared to placebo, on the change in concentration of inflammatory cytokines in blood.
Number of abnormal clinically significant findings (physical, neurological, ophthalmological and dermatological examinations). | Up to 6 weeks
Number of abnormal clinically significant findings in clinical laboratory assessments (hematology, coagulation, clinical chemistry, urinalysis). | Up to 6 weeks
Number of abnormal clinically significant findings in electrocardiogram results. | Up to 6 weeks
  The following electrocardiogram parameters will be assess: PR interval, QRS interval, RR interval, QT interval and QTc interval.
Number of abnormal clinically significant findings in vital signs assessments (respiratory, body temperature, blood pressure, pulse). | Up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (16):
- Poland (2):
  - Mazowiecki Szpital Bródnowski, Warsaw, Masovian Voivodeship
  - Instytut Zdrowia dr Boczarska-Jedynak Sp. Z o.o., Sp. K.,, Oświęcim, Małopolska
- Ukraine (14):
  - Cherkasy Regional Hospital of the Cherkasy Regional Council, Cherkasy
  - Ukrainian State Research Institute of Medical and Social Problems of Disability of the Ministry of Health of Ukraine, Department of Neurology and Borderline Conditions;, Dnipro
  - Treatment and Diagnostic Centre "Neuro Global" of the Limited Liability Company "Neuro Global", Treatment and Prevention Sub-division, Ivano-Frankivsk
  - Institute of Neurology, Psychiatry and Narcology of the Academy of Medical Sciences of Ukraine, Department of Vascular Pathology of the Brain and Rehabilitation, Kharkiv
  - "Medical center "Dobrobut-Polyclinic" "Medical diagnostic center "Dobrobut", Kyiv
  - Medical Center of the Limited Liability Company "Medical Center "Consilium Medical", Kyiv
  - "D.F. Chebotaryov Institute of Gerontology of the National Academy of Medical Sciences of Ukraine, Kyiv
  - Municipal non-profit enterprise of Lviv regional council "Lviv regional clinical hospital", Neurological Department, Lviv
  - Poltava Regional Clinical Hospital named after M.V. Sklifosovsky of the Poltava Regional Council, Poltava
  - Limited Liability Company, Medical Center "DIAMED", Uzhhorod
  - Medical Center of the Limited Liability Company "Salyutem Medical Center", Vinnytsy
  - "INET-09" LLC (Medical Center), Zaporizhzhia
  - Educational and Scientific Medical Center "University Clinic" of Zaporizhzhia State Medical University, Zaporizhzhia
  - Communal Enterprise "Hospital" of Zhytomyr City Council, Zhytomyr